CLINICAL TRIAL: NCT02612753
Title: Interest of Combining Speech Therapy With a Non-invasive Brain Stimulation (tDCS) for the Aphasic Patient
Acronym: Taph
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Paul Bennetot (Other); Fondation Garches (Other)
Responsible Party: Principal Investigator, AZOUVI, MDPHD, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-A01773-44
Record Dates: First submitted 2015-10-29; First posted 2015-11-24 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Aphasia
Keywords: Aphasia; Speaking therapy; Language therapy; transcranial Direct current stimulation
MeSH Terms: conditions — Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aphasics Patients (Experimental): Patients which have difficulties to speak. Improvement of language for aphasics patients.
  Interventions: Procedure: improvement of language for aphasics patients; Device: tDCs
- Aphasics Patients control (Sham Comparator): Patients which have difficulties to speak will receive Sham tDCS +SLT for aphasics patients control
  Interventions: Procedure: improvement of language for aphasics patients; Device: Sham tDCS

INTERVENTIONS:
Procedure: improvement of language for aphasics patients — Aphasics patients receive active stimulation during SLT
Device: Sham tDCS — Aphasics patients control receive sham stimulation during SLT
  Arms: Aphasics Patients control
Device: tDCs
  Arms: Aphasics Patients

SUMMARY:
Aphasia is a frequent symptom after a left hemisphere stroke. It has serious impacts on social, family and professional lives. Aphasic patients need to be rehabilitated. To date, no pharmacological treatment being available only speech and language therapy (SLT) can improve patients, but its efficiency is moderate. Several studies have investigated the link between the recovery of language and neural reorganization. tDCs, a noninvasive technology for modulating neural excitability, could potentiate the effects of the SLT. About 25 studies in literature have described beneficial effects of tDCs coupled with SLT on aphasic patients. However to the investigator knowledge the feasibility of tDCs and speech therapy in clinical pathways has never been investigated. That is why the investigator propose to study in real care conditions how SLT proves more efficient on the recovery of language in a discursive assessment when coupled with active stimulation than with placebo stimulation.

DETAILED DESCRIPTION:
This is a multicenter, cross-over, randomized, controlled and double blind study. 24 patients will be included between November 2015 and November 2017.

During each session of speech and language treatment, aphasics will receive a weak 2 milli amperes (electric) current delivered by a tDCs device for 20 minutes. The stimulation will be either active or placebo. Each stage of the cross over will last three weeks. Patients will be administered the usual number of SLT sessions, no particular therapy being imposed. To evaluate the long-time effects of the therapy, three follow-up measures will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years
* Aphasic Following a brain injury identified by MRI.
* Present a aphasia severity score> 1 on the Boston Diagnostic Aphasia Examination (BDAE) severity scale.
* No Post stroke delay is retained but the patient should be stable from a medical point of view.
* Master Of the French language in spoken and written
* Affiliated to a social security
* Patient Who signed the informed consent

Exclusion Criteria:

* Other previous neurological pathologies
* epileptic crisis during the previous 2 months
* Patient denies
* Presence of a cranial flap
* intracerebral metal hardware Presence
* Patient under guardianship
* Patient unable to understand the study
* Patient subject to an exclusion period for another search.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
change of number of names, without error and not repeated in the speech | Baseline measures: start of Week 1, 2 and 3. Outcomes measures: 1 assessment at the end of the 5 th week, 1 at the beginning of the 7th week, 1 at the end of the 9 th week and 1 at the end of the 10th week. Follow-up measures: 12th, 14th, 16th
  The participant must answer a simple question "explain me your job or your study". Their production will be recorded and analyzed.
  For evaluate the stability of participant performances before the stimulation period three based line will be propose. The third base line corresponds to the start of the first stimulation period. After the three week of tdcs coupled with the SLT a new assessment will be realized. One week later begin the new stage of cross over. An assessment will be administered just before and just after the second stimulation period. Then, three follow-up assessments (one all two weeks) will be proposed during one and half month.

SECONDARY OUTCOMES:
verbal fluency | Baseline measures: start of Week 1, 2 and 3. Outcomes measures: 1 assessment at the end of the 5 th week, 1 at the beginning of the 7th week, 1 at the end of the 9 th week and 1 at the end of the 10th week. Follow-up measures: 12th, 14th, 16th week.
  the participant has two minutes to find the most animal names words beginning by letter p. Investigator collect the number of correct words and calculate the standard deviation according to published norms.
working memory | baseline measures: start of Week 1, 2 and 3. Outcomes measures: 1 assessment at the end of the 5 th week, 1 at the beginning of the 7th week, 1 at the end of the 9 th week and 1 at the end of the 10th week. Follow-up measures: 12th, 14th, 16th week.
  the participant repeats the numbers in the same order or inverted order. Investigator collect the highest group of number repeated
visual exploration | baseline measures: start of Week 1, 2 and 3. Outcomes measures: 1 assessment at the end of the 5 th week, 1 at the beginning of the 7th week, 1 at the end of the 9 th week and 1 at the end of the 10th week. Follow-up measures: 12th, 14th, 16th week.
  a paper with a lot of drawing is presented to the participant. The participant must delete all the bells as fast as possible. Investigator collect the number of bell omissions
every day life scale | Baseline measures: start of Week 1, 2 and 3. Outcomes measures: 1 assessment at the end of the 5 th week, 1 at the beginning of the 7th week, 1 at the end of the 9 th week and 1 at the end of the 10th week. Follow-up measures: 12th, 14th, 16th week.
  a questionnaire is proposed to the participant in order to better understanding how is the communication with their close or with unknown person in a conversation or phone
likert scale | at the end of the 9 th week, a likert 5 grade scale was proposed.
  likert scale are proposed to know how the stimulation is tolerated and accepted by the participant, the patient family and the speech therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe AZOUVI, MDPHD, Principal Investigator — Hopital RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France

REFERENCES:
- [Result] Greener J, Enderby P, Whurr R. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2000;(2):CD000425. doi: 10.1002/14651858.CD000425. PMID 10796360
- [Result] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Result] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving aphasia in patients with aphasia after stroke. Cochrane Database Syst Rev. 2015 May 1;(5):CD009760. doi: 10.1002/14651858.CD009760.pub3. PMID 25929694
- [Result] Robey RR. A meta-analysis of clinical outcomes in the treatment of aphasia. J Speech Lang Hear Res. 1998 Feb;41(1):172-87. doi: 10.1044/jslhr.4101.172. PMID 9493743
- [Result] Klippi A, Sellman J, Heikkinen P, Laine M. Current clinical practices in Aphasia Therapy in Finland: challenges in moving towards national best practice. Folia Phoniatr Logop. 2012;64(4):169-78. doi: 10.1159/000341106. Epub 2012 Oct 25. PMID 23108446